CLINICAL TRIAL: NCT04469556
Title: Pancreatic Adenocarcinoma Signature Stratification for Treatment
Acronym: PASS-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Johns Hopkins University (Other); Cold Spring Harbor Laboratory (Other); Ontario Institute for Cancer Research (Other); Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASS-01; CAPCR ID: 20-5105 (Other: UHN)
Record Dates: First submitted 2020-06-26; First posted 2020-07-14 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Ductal Adenocarcinoma; Advanced Pancreatic Cancer
MeSH Terms: interventions — folfirinox; Irinotecan; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Approximately 150 patients will be randomized in a 1:1 ratio to receive one of the two standard of care regimens in patients with confirmed metastatic PDAC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Folfirinox (Active Comparator): Modified FOLFIRINOX (Folinic acid/Leucovorin, 5-Fluouracil, Irinotecan, Oxaliplatin) administered intravenously.
  Given that both regimens are standard of care, study treatment will be administered as per standard of care at each institution including a maintenance therapy approach which is encouraged in both arms. Dose modifications, anti-emetics, supportive medications, and use of growth factors should follow institutional guidelines.
  Interventions: Drug: Folfirinox
- Gemcitabine/nab-Paclitaxel (Active Comparator): Gemcitabine/nab-Paclitaxel administered intravenously.
  Given that both regimens are standard of care, study treatment will be administered as per standard of care at each institution including a maintenance therapy approach which is encouraged in both arms. Dose modifications, anti-emetics, supportive medications, and use of growth factors should follow institutional guidelines.
  Interventions: Drug: Gemcitabine/nab-paclitaxel

INTERVENTIONS:
Drug: Folfirinox — Chemotherapy
  Other Names: Folinic Acid/Leucovorin, 5-Fluouracil, Irinotecan, Oxaliplatin
  Arms: Modified Folfirinox
Drug: Gemcitabine/nab-paclitaxel — Chemotherapy
  Arms: Gemcitabine/nab-Paclitaxel

SUMMARY:
This is a randomized multicentre phase II trial with a large translational component. The trial will evaluate the two standard chemotherapy regimens: modified folfirinox (mFFX) and gemcitabine/nab-paclitaxel (GA), in patients with untreated metastatic pancreatic ductal adenocarcinoma. Integrated into this phase II trial are a number of laboratory components including molecular profiling, patient derived organoid establishment, and drug testing sensitivity and other biomarkers.

DETAILED DESCRIPTION:
The two chemotherapy regimens GA and mFFX remain standard treatment options without biomarkers to predict response. PASS-01 will for the first time explore progression free survival differences in the two standard backbone regimens used in the advanced setting. Biomarker driven strategies in pancreatic ductal adenocarcinoma (PDAC) are lacking, perhaps accounting for a large number of failed phase II studies. This study will evaluate two standard of care chemotherapy regimens, but will also explore high content molecular profiling, chemotherapy sensitivity signatures, GATA6 and other putative biomarkers as predictors of response to chemotherapy. In addition, the use of patient derived organoid models for personalized medicine in PDAC will continue to develop within this study.

Approximately 150 patients diagnosed with untreated metastatic pancreatic cancer will be randomized to either arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histological or radiological diagnosis of untreated metastatic PDAC at screening with histology subsequently confirmed prior to randomization.
2. Eligible histologic variants include adenocarcinoma or variants to include mucinous adenocarcinoma or adenosquamous carcinoma.
3. Patients with a history of prior or concurrent second primary malignancy whose natural history or treatment does not have the potential to interfere with the safety or primary endpoint efficacy assessment of the pancreas cancer should generally be eligible for enrollment in clinical trials.
4. Age ≥18 years.
5. Patient must have a tumor lesion that is amenable to a core needle biopsy.
6. Patients must be suitable for treatment with either mFFX and GA without contraindications to either regimen.
7. Eastern Cooperative Group (ECOG) performance status 0-1. (Karnofsky ≥70%).
8. Life expectancy of greater than 90 days, as judged by the investigator
9. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test and must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
10. Within 14 days of the proposed randomization date, patients must have normal organ and marrow function

Exclusion Criteria:

1. Patients who have received prior systemic treatment for PDAC, including treatment in the neoadjuvant or adjuvant setting. Prior surgery or palliative radiation is permitted.
2. Patients with histology other than pancreatic ductal adenocarcinoma. Those with adenosquamous are allowed. Acinar tumors and colloid are excluded.
3. Patients with one or more contraindications to tumor biopsy according to local institution's standard biopsy procedures.
4. Patients with known brain metastases are excluded from participation in this clinical study.
5. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, inability to stop anticoagulation medication for a biopsy, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
7. Patients with a known germline mutation in BRCA, PALB2 or other homologous Recombination Repair Deficiency (HRD) genes.
8. Patients who are pregnant or breastfeeding.
9. Use (including 'recreational use') of any illicit drugs or other substance abuse (including alcohol) that could potentially interfere with adherence to study procedures or requirements. *Use of any illicit drugs or other substance abuse (including alcohol) are not screened in Canada using Toxicity testing. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) in mFFX and GA arms pancreatic ductal adenocarcinoma (PDAC) in a randomized phase II trial. | 2-4 years
  Time from the date of randomization to progression based on the radiology assessment of response using RECIST v1.1, or death, whichever is earlier

SECONDARY OUTCOMES:
ORR by RECIST 1.1 and duration of response in patients receiving mFFX or GA | 2-4 years
  percentage of patient's measurable disease who have achieved either complete response (CR) or partial response (PR)
Overall survival (OS) associated with mFFX or GA profiles, signatures and pharmacotyping | 2-4 years
GATA6 as a biomarker of response to mFFX or GA | 2-4 years
• Concordance between organoid transcriptomic profiles (RNAseq) and patient transcriptomic profiles (descriptive statistics) | 2-4 years
• Concordance between chemotherapy sensitivity signature predictions and response to first line treatment (descriptive statistics). | 2-4 years
• Correlation of individual tumour cytokeratins (eg. CK5 and CK17 expression) with chemotherapy response and resistance | 2-4 years
Cell free circulating tumor (ct) DNA analysis (including KRAS mutational status) | 2-4 years
Cluster Tendency analysis using artificial neural networks and radiomic methods combined | 2-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jaffee, MD, Study Chair — Johns Hopkins University; Jennifer J Knox, MD, Study Chair — University Health Network, Toronto
Locations (6):
- United States (4):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Northwell Health, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Canada (2):
  - BC Cancer Agency Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No